CLINICAL TRIAL: NCT01661842
Title: Phase 1/2 Study of UC-MSC Treatment for Evaluation the Efficacy and Safety in Patients With Autoimmune Liver Disease
Brief Title: Umbilical Cord Mesenchymal Stem Cells for Patients With Autoimmune Hepatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Director of both the Research Center for Biological Therapy and the Beijing Institute of Translational Hepatology, Beijing 302 Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302-006
Record Dates: First submitted 2012-08-05; First posted 2012-08-10 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune Hepatitis; Mesenchymal stem cells; serum albumin; serum Tbil; serum immunoglobulin G(IgG)
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional plus UC-MSC treatment (Experimental): Participants will receive conventional treatment plus a dose of UC-MSC from day 0 through the week 12 study visit.
  Participants will then be followed until the week 96 study visit.
  Interventions: Other: conventional plus UC-MSC treatment
- Conventional plus placebo treatment (Experimental): Participants will receive conventional plus placebo treatment from day 0 through the week 12 study visit. Participants will then be followed until the week 96 study visit.
  Interventions: Other: Conventional plus placebo treatment

INTERVENTIONS:
Other: conventional plus UC-MSC treatment — Received conventional treatment and taken i.v., once per 4 week, at a dose of 1×106 UC-MSC/kg body weight for 12 weeks.
  Arms: Conventional plus UC-MSC treatment
Other: Conventional plus placebo treatment — Received conventional treatment and taken i.v., once per 4 week, at 50 ml saline for 12 weeks
  Arms: Conventional plus placebo treatment

SUMMARY:
Autoimmune hepatitis (AIH) is characterized by chronic inflammation of the liver, interface hepatitis, hypergammaglobulinemia, and the presence of autoantibodies. Disease presentation is varied but typically is based on characteristic aminotransferase elevations, histological abnormalities, elevated levels of serum globulins, and the presence of one or more autoantibodies. Two types of juvenile AIH have been identified according to seropositivity for smooth muscle and /or antinuclear antibody (AIH type 1) or liver kidney microsomal antibody (AIH type 2). Standard therapy in clinic consists of a combination of corticosteroids and azathioprine, which displays the efficacy in 80% of patients. However, 7% of patients deteriorate despite compliance with the standard corticosteroid regiments (treatment failure),13% of patients improve but not to a degree that satisfies remission criteria (incomplete response), 13% of patients develop serious drug-induced complications, and 50%-86% of patients will relapse after drug withdrawal. These serious drawbacks counterbalance the benefits of conventional therapy, and they are compelling reasons to refine current treatment strategies and pursue alternative therapies. UC-MSC has been the application for the treatment of several severe autoimmune diseases, such as immune thrombocytopenia, systemic lupus erythematosus, and therapy-resistant rheumatoid arthritis. In this study, the safety and efficacy of UC-MSC transplantation for AIH patients will be evaluated.

DETAILED DESCRIPTION:
Autoimmune hepatitis (AIH) is an immune-mediated necroinflammatory disease of the liver characterized by elevation of IgG, presence of characteristic autoantibodies, and histological feature of interface hepatitis. Standard therapy consists of a combination of corticosteroids and azathioprine, which is efficacious in 80% of patients. However, current treatment strategies are complicated by frequent relapse after drug withdrawal, medication intolerance, and refractory disease. Alternative medical therapy may be need for AIH.

The potential for stem cells to differentiate into hepatocytes cells was recently confirmed. In particular, bone marrow-derived mesenchymal stem cell (BM-MSC) transplantation has been applicated in the clinic for treat several human disease such as GVHD, cardiac injury and brain injury, and displayed good tolerance and efficiency. Recently, umbilical cord-derived MSCs (UC-MSC) has also been used to treat severe autoimmune diseases, such as immune thrombocytopenia, systemic lupus erythematosus, and therapy-resistant rheumatoid arthritis.

The purpose of this study is to learn whether and how UC-MSC can improve the disease condition in patients with autoimmune hepatitis (AIH). This study will also look at how well UC-MSC is tolerated and its safety in AIH patients

Participants in the study will be randomly assigned to one of two treatment arms:

Arm A: Participants will receive 12 weeks of UC-MSC treatment plus conventional treatment (combination of corticosteroids and azathioprine) Arm B: Participants will receive 12 weeks of placebo plus conventional treatment. (combination of corticosteroids and azathioprine) UC-MSC will be prepared according to standard procedures and is collected in plastic bags containing anticoagulant. UC-MSCs are given via i.v. under sonography monitoring. After cell therapy, patients are followed up at week 12, 24, 36, 48, 72, 96. The evaluation of some clinical parameters such as the level of serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), γ-globulin, total bilirubin (TB), prothrombin time (PT), albumin (ALB), prealbumin (PA) and IgG, are detected at these time points. MELD score, Liver histology, treatment side effects, relapse rate and clinical symptoms were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Autoimmune hepatitis (according to the criteria defined by the international autoimmune hepatitis Group ,Hepatology, 2008;48:169-176)
3. Negative pregnancy test (female patients in fertile age)

Exclusion Criteria:

1. Hepatocellular carcinoma or other Malignancies
2. Pregnant or lactating women
3. Viral Hepatitis ( HAV,HBV,HCV, et al )
4. Vital organs failure (Cardiac, Renal or Respiratory, et al)
5. Sepsis
6. Active thrombosis in the portal or hepatic veins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Liver Histology change | baseline and 96 weeks
Serum alanine aminotransferase (ALT) | 0,12, 24, 36, 48, 72, 96 weeks after treatment

SECONDARY OUTCOMES:
Serum AST | At baseline and at week 12, 24, 36, 48, 72, 96
Serum Tbil | At baseline and at week 12, 24, 36, 48, 72, 96
Serum immunoglobulin G (IgG) | At baseline and at week 12, 24, 36, 48, 72, 96
Serum γ-globulin | At baseline and at week 12, 24, 36, 48, 72, 96
MELD score | At base line and at week 12, 24, 36, 48, 72, 96
Number of participants with treatment side effects | At base line and at week 12, 24, 36, 48, 72, 96
  weight gain, acne, facial rounding, dorsal hump formation, hirsutism, osteopenia and diabetes mellitus, et al
Number of participants with improvement of clinical symptoms | At base line and at week 12, 24, 36, 48, 72, 96
  diffuse arthralgias, fatigue, generalized malaise, jaundice, abdominal pain, nausea, and loss of appetite

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, professor, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Czaja AJ. Advances in the current treatment of autoimmune hepatitis. Dig Dis Sci. 2012 Aug;57(8):1996-2010. doi: 10.1007/s10620-012-2151-2. Epub 2012 Apr 3. PMID 22476586
- [Background] Montano-Loza AJ, Carpenter HA, Czaja AJ. Features associated with treatment failure in type 1 autoimmune hepatitis and predictive value of the model of end-stage liver disease. Hepatology. 2007 Oct;46(4):1138-45. doi: 10.1002/hep.21787. PMID 17668882
- [Background] Czaja AJ. Promising pharmacological, molecular and cellular treatments of autoimmune hepatitis. Curr Pharm Des. 2011;17(29):3120-40. doi: 10.2174/138161211798157568. PMID 21902661
- [Background] Gossard AA, Lindor KD. Autoimmune hepatitis: a review. J Gastroenterol. 2012 May;47(5):498-503. doi: 10.1007/s00535-012-0586-z. Epub 2012 Apr 17. PMID 22526272
- [Background] Malekzadeh Z, Haghazali S, Sepanlou SG, Vahedi H, Merat S, Sotoudeh M, Nasseri-Moghaddam S, Malekzadeh R. Clinical features and long term outcome of 102 treated autoimmune hepatitis patients. Hepat Mon. 2012 Feb;12(2):92-9. doi: 10.5812/hepatmon.808. Epub 2012 Feb 29. PMID 22509185
- [Background] Yi T, Song SU. Immunomodulatory properties of mesenchymal stem cells and their therapeutic applications. Arch Pharm Res. 2012 Feb;35(2):213-21. doi: 10.1007/s12272-012-0202-z. Epub 2012 Feb 28. PMID 22370776
- [Background] Holbro A, Abinun M, Daikeler T. Management of autoimmune diseases after haematopoietic stem cell transplantation. Br J Haematol. 2012 May;157(3):281-90. doi: 10.1111/j.1365-2141.2012.09070.x. Epub 2012 Feb 24. PMID 22360687